CLINICAL TRIAL: NCT02361788
Title: A Prospective Cohort Study on the Etiology of Neonatal Hyperbilirubinemia in a Migrant and Refugee Population on the Thai-Myanmar Border
Brief Title: Study on Newborn Babies With a Yellow Skin Color (Neonatal Jaundice Study)
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU 1307
Record Dates: First submitted 2014-09-01; First posted 2015-02-12 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2022-07

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: neonatal hyperbilirubinemia; etiology; incidence; risk factors
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Neonatal hyperbilirubinemia is the most common reason for admission in the neonatal period (first month of life) worldwide and at SMRU. The skin of the newborn baby becomes jaundiced, which is caused by a high level of bilirubin in the blood. In some neonates the level of bilirubin increases to a level that can cause braindamage or even death. There are different causes known that can lead to higher levels of bilirubin, for example G6PD deficiency and prematurity. In case of neonatal hyperbilirubinemia the neonate needs to be treated with phototherapy (blue light therapy). If there is prolonged jaundice (≥ 21 days), further investigations needs to be done.

Objectives:

Primary objective:

To determine the etiology of neonatal hyperbilirubinemia in neonates with a gestational age of ≥ 28 weeks from the refugee and migrant population, on the Thai-Myanmar border.

Secondary objective:

* Establishing the incidence of neonatal hyperbilirubinemia
* Determine the risk factors for the development of neonatal hyperbilirubinemia
* Determine the incidence of prolonged neonatal jaundice
* Determine the neurodevelopmental outcome, at the age of 6 and 12 months
* Determine the body composition, using air-displacement plethysmography, at birth, 1, 2 and 3 months of age
* Determine the incidence of anaemia and illness episodes during the first year of life
* Determine the incidence of helminthic infection at the age of one year
* Assess the knowledge level and misbeliefs on neonatal hyperbilirubinemia among the mothers and SMRU health care staff

Research design: The study will conduct an exhaustive prospective descriptive study, all eligible newborns will be enrolled after obtaining the informed consent from their mothers. During pregnancy and delivery we will collect clinical data about the mother. At birth we will take umbilical cord blood (9 ml) to test for different causes of neonatal hyperbilirubinemia. In the first week of life we plan 4 moments to measure the bilirubin and hematocrit level (0.05 ml), weight and ask questions about feeding and other practices. Based on the bilirubin results we will determine whether the neonate needs phototherapy. After the first week we weekly follow-up will be conducted and in case of visible jaundice we will measure the bilirubin level. If the neonate is still jaundiced after the age of 21 days we will further investigate the cause. In the infant period, until the age of one year, we plan to have monthly follow-up to assess the health and growth of the child and at the age of 3, 6 and 12 months we will do a neurodevelopmental test.

An improved understanding of the pathological processes contributing to the development of neonatal hyperbilirubinemia is needed in order to to identify neonates at risk and develop improved management.

DETAILED DESCRIPTION:
PROCEDURES DURING PREGNANCY

During the first antenatal care visit the mother will have a gestational dating ultrasound to determine the accurate gestational age. During all antenatal care visits information about the mother will be collected as part of standard obstetric care:

* Ethnicity
* Age
* Medical history

  * Blood transfusion in history
  * Chronic diseases
* Obstetric history

  * Parity and gravida
  * Previous neonatal deaths and reason of death
  * Previous preterm delivery
  * Previous child with neonatal hyperbilirubinemia
* Pregnancy

  * Gestational dating ultrasound
  * Obstetric problems
  * Malaria and morbidity episodes during pregnancy
  * BMI, MUAC and weightgain
  * Laboratory results

    * Hepatitis B status*
    * HIV status*
    * Syphilis serology*
    * G6PD status
    * Hemoglobinopathy
    * ABO blood group
    * Rhesus D blood group

Testing for STD and HIV is routine practice at the SMRU clinics. Before the screening permission from the mother is requested. Life-long antiretroviral triple therapy is available in case of a positive HIV test.

To assess the knowledge and beliefs on neonatal jaundice among the mothers we will perform a short questionnaire. This questionnaire will help the study team to assess the level of knowledge and the misbeliefs on neonatal hyperbilirubinemia. The study team will also ask the subjects about the use of naphthalene containing moth balls and explain them the danger in case the subject's baby will be G6PD deficient.

PROCEDURES AT BIRTH

Eligibility:

At birth the neonate will be excluded if the gestational age is < 28 weeks.

Questionnaire:

Detailed data about the delivery will be collected:

* Duration of maternal membrane rupture before delivery
* Mode of delivery
* Presence of maternal fever in labour and use of antibiotics
* Use of oxytocin
* Complications
* Gestational age

  * Confirmed by ultrasound if presenting < 24 weeks (CRL < 14 weeks, HC 14-23+6) or, in case of late ultrasound, determined with the Dubowitz gestational age assessment (performed 6-72 hours after birth)
* Apgar score and need for resuscitation
* Gender

Laboratory Investigations:

Umbilical cord blood will be obtained for laboratory investigations as below;

ABO and Rhesus D blood group 0.1 ml., G6PD fluorescent test 0.005 ml., G6PD spectrophotometric assay 0.05 ml., G6PD flow cytometric assay 0.05 ml., Coomb's test (Direct Antiglobulin Test) 3 ml., Albumin 3 ml., Genotyping (G6PD, SAO, UGT1A1 mutations) 2 ml.,

Total volume 8.205 ml (For practical reason we will take 9 ml.)

Clinical assessment:

Birthweight, length and head circumference will be determined. The body composition will be measured using air-displacement plethysmography (PeaPod) . A newborn physical examination (including vital signs) will be performed within the first 24 hours, as part of normal neonatal care:

Observations:

* skin colour (pale/cyanosed/jaundiced/normal),
* skin rash
* description of anterior fontanelle (raised/normal/depressed),
* bruising on the body: location
* swelling on the head

  * 2 diameters will be measured
  * swelling crossing the scalp sutures
  * diagnose: caput succedaneum, cephalhematoma or subgaleal hemorrhage
* abnormality of the face
* abnormality of palate, mouth
* abnormality of limbs, fingers or toes

Cardiovascular examination: heart rate(per minute), heart sounds, femoral pulses

Respiratory examination: respiratory rate (per minute), lung sounds, signs of respiratory distress (chest indrawing/nasal flaring/head bobbing)

Abdominal examination: abdominal mass, enlarged liver or spleen, genitalia, anus

Neurological examination: muscle tone, moving of limbs, eye red reflex

PROCEDURES DURING NEONATAL FOLLOW-UP In the first week after birth there are four moments when the neonate will be assessed. This will be 24 hours [range 22-26 hours], 48 hours [range 36-60 hours], 84 hours [range 70-96 hours] and on day 6 [range day 5-8]. After this week the mother will be asked to come back for weekly follow-up until the age of one month. At one month of age the body composition will be measured using PeaPod.

Questionnaire:

The mother will be asked questions:

First 24 hours after delivery:

* Age (in hours) of initiation of feeding
* Feeding:

  * How is the baby being fed (exclusive breastmilk, supplementary or mixed feeding)
  * If supplementary feeding, what is the reason for this?
  * Does the baby suck well?
* Use of drugs or herbal medicine by mother in first 24 hours
* Use of herbal preparations for neonate
* Age (in hours) at passage of first stool and urine
* Use of napthalene balls for storing of baby clothes

During every follow-up the mother the questions about feeding will be repeated.

Laboratory Investigations:

During every neonatal follow-up until the visit on day 6 [range day 5-8], a SBR and haematocrit will be measured. The SBR result will be plotted, by age on a jaundice treatment graph specific for the gestational age and the need for phototherapy or more intense follow-up will be determined. During weekly follow-up after the age of 8 days, only a SBR and hematocrit will be measured in case of visible jaundice. At the age of one month, a hematocrit will be measured for anemia screening and the G6PD fluorescent test will be repeated as below.

Serum bilirubin 0.05 ml. x 5, Haematocrit 0.05 ml. x 5, G6PD fluorescent test 0.005 ml.

Total 0.205 ml.

Clinical assessment:

A physical examination (including vital signs) will be performed at every visit and the weight will be measured. Weightloss or -increase will be calculated and if there is ≥ 10% weightloss, the neonate will be reviewed carefully for any underlying cause of this weightloss and supplementary feeding (expressed breastmilk or powdermilk) will be started.

PROCEDURES WHEN DELIVERY OUTSIDE SMRU

In case of delivery in another clinic or at home, but the mother and neonate visit a SMRU clinic within the first 48 hours after delivery, the neonate can still be included in the study.

If a neonate is born outside SMRU and does not visit the clinic within 48 hours after delivery, but presents with neonatal hyperbilirubinemia in the first 8 days of life, this neonate can be included in the study as well. Because no umbilical cord blood was taken, a limited set of laboratory investigations will be performed, as described as below;.

ABO and Rhesus D bloodgroup 0.075 ml., G6PD fluorescent test 0.005 ml., G6PD spectrophotometric assay 0.05 ml., G6PD flow cytometric assay 0.05 ml., Serum bilirubin 0.05 ml., Haematocrit 0.05 ml., Genotyping 2 ml.,

Total volume 2.23 ml.

PROCEDURES DURING INFANT FOLLOW-UP

Infant follow-up will take place every month until the age of 12 months.

Questionnaire:

At every visit the mother will be asked about feeding practices and after the age of 6 months about neurodevelopmental milestones.

Laboratory investigations:

Due to the problems of anaemia in this population (50% of the infants are reported to have a haematocrit of < 33% at the age of 6 months; personal communication Dr. Rose McGready) haematocrit will be measured monthly, by finger prick, and anaemia will be treated if necessary. At the age of one year a stool test for parasitology screening will be taken and the infant will be treated if necessary. Finally at one year of age the infant will be screened for hemoglobinopathy due to contradictory reports of the association between neonatal hyperbilirubinemia and hemoglobinopathy as below:

Haematocrit 0.05 ml. x11, Hemoglobin typing 3 ml.

Total volume 3.55 ml.

Clinical assessment:

A physical examination (including vital signs) will be performed at every visit and the weight will be measured. At the age of 2 and 3 month a body composition will be measured using PeaPod. At 3, 6, 9 and 12 months the length and head circumference will be measured.

At the age of 3, 6 months and 12 months the infant will be assessed with the Shoklo Developmental Test 53 and the results compared to age specific norms developed for this population.

Funder & grant reference number: This research was funded in whole, or in part, by the Wellcome Trust [grant 220211]. For the purpose of Open Access, the authors have applied a CC BY public copyright license to any author accepted manuscript version arising from this submission. LT was supported by a PhD grant from "The Belgian Kids Fund for Pediatric Research:2017-2018".

Summary of results:

Population risks for neonatal hyperbilirubinaemia (NH) vary. Knowledge of local risks permits interventions that may reduce the proportion becoming severe. Between January 2015 and May 2016, in a resource-limited setting on the Thailand-Myanmar border, neonates from 28 weeks' gestation were enrolled into a prospective birth cohort. Each neonate had total serum bilirubin measurements: scheduled (24, 48, 72 and 144 hours of life) and clinically indicated; and weekly follow up until 1 month of age. Risk factors for developing NH were evaluated using Cox proportional hazard mixed model. Of 1710 neonates, 22% (376) developed NH (83% preterm, 19% term). All neonates born <35 weeks, four in five born 35- 37 weeks, and three in twenty born >38 weeks had NH, giving an overall incidence of 249 per 1000 livebirths [95%CI 225, 403]. Mortality from acute bilirubin encephalopathy was 10% (2/20) amongst the 5.3% (20/376) who reached the severe NH threshold. One-quarter (26.3%) of NH occurred within 24 hours. NH onset varied with gestational age: at a median [IQR] 24 hours [24, 30] for neonates born 37 weeks or prematurely vs 59 hours [48, 84] for neonates born >38 weeks. Risk factors for NH in the first week of life independent of gestational age were: neonatal G6PD deficiency, birth bruising, Sgaw Karen ethnicity, primigravidae, pre-eclampsia, and prolonged rupture of membranes. The genetic impact of G6PD deficiency on NH was partially interpreted by using the florescent spot test and further genotyping work is in progress. The risk of NH in Sgaw Karen refugees may be overlooked internationally as they are most likely regarded as Burmese in countries of resettlement. Given high levels of pathological jaundice in the first 24 hours and overall high NH burden, guidelines changes were implemented including preventive PT for all neonates <35 weeks and for those 35-37 weeks with risk factors.

FST was performed on 1521 umbilical cord blood samples. Quality control and genotyping revealed 10 misdiagnoses. After quality control, 10.7% of the males (84/786) and 1.2% of the females (9/735) were phenotypically G6PD deficient at birth. The FST repeated at one month of age or later diagnosed 8 additional G6PD deficient infants who were phenotypically normal at birth.

Lower gestational age (<38 weeks), mutations in the genes encoding glucose-6-phosphate dehydrogenase (G6PD) and uridine 50-diphospho-glucuronosyltransferase (UGT) 1A1 were identified as the main independent risk factors for NH in the first week, and for prolonged jaundice in the first month of life. Population attributable risks (PAR%) were 61.7% for lower gestational age, 22.9% for hemi or homozygous and 9.9% for heterozygous G6PD deficiency respectively, and 6.3% for UGT1A1*6 homozygosity. In neonates with an estimated gestational age ≤38 weeks, G6PD mutations contributed PARs of 38.1% and 23.6% for "early" (≤48 hours) and "late" (49-168 hours) NH respectively. For late NH, the PAR for UGT1A1*6 homozygosity was 7.7%. Maternal excess weight was also a significant risk factor for "early" NH while maternal mutations on the beta-globin gene, prolonged rupture of membranes, large haematomas and neonatal sepsis were risk factors for "late" NH. For prolonged jaundice during the first month of life, G6PD mutations and UGT1A1*6 mutation, together with lower gestational age at birth and presence of haematoma were significant risk factors.

Conclusions:

In this resource-limited setting with a dedicated special baby care unit but not intensive care nor timely access to exchange transfusion, this epidemiological study identified a high NH prevalence, 1 in 4 developing within 24 hours of life. Active screening likely lowered severe case incidence but mortality due to encephalopathy was still 1 in 10, and this is probably an underestimate. Guidelines were modified towards early NH identification and treatment and adequate follow up of those at risk of late NH. Sgaw Karen have the highest risk of NH according to ethnicity but are internationally known as Burmese refugees. The increased risk of NH in neonates identified as G6PD deficient by fluorescent spot test most likely underestimate the risk in female neonates and further research is currently evaluating this. This study demonstrates that mortality and potentially crippling morbidity from severe NH can be managed in a resource limited setting that can provide screening for TSB and offer phototherapy based on guidelines.

This study shows the short-comings of the G6PD FST in neonatal routine screening and highlights the importance of training and quality control.

In this population, genetic factors contribute considerably to the high risk of NH. Diagnostic tools to identify G6PD deficiency quantitatively at birth would facilitate early recognition of high risk cases.

ELIGIBILITY:
Inclusion Criteria:

* Written or thumb print informed consent from the mother during pregnancy
* Neonates who are born to mothers who followed antenatal care at SMRU antenatal clinics
* Neonates who are born in a SMRU clinic OR neonates who are born outside SMRU but visit a SMRU clinic within 48 hours after birth OR neonates who are born outside SMRU and present with neonatal jaundice at any moment in the first 8 days

Exclusion Criteria:

* No written or thumb print informed consent from the mother during pregnancy
* Neonates who are born to mothers who did not follow antenatal care
* Neonates < 28 weeks gestation
* Neonate born outside SMRU and present > 48 hours after delivery without jaundice

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Over the course of a one year period, the mothers of neonates (estimated gestation ≥ 28 weeks) who meet the inclusion criteria and none of the exclusion criteria will be asked to participate in this study.
  Based on previous experience, assuming that most mothers will agree to participate in the study and 15% of the included neonates will be lost before completion of the study, we will include approximately 1887 neonates. With an estimated proportion of neonatal hyperbilirubinemia of 18%, 340 of 1887 neonates will develop neonatal hyperbilirubinemia. Other prospective studies had numbers of neonates with neonatal hyperbilirubinemia ranging from 21 to 624.
Sampling Method: Non-Probability Sample
Enrollment: 1710 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2016-06-12 (Actual); Study Completion 2019-05-18 (Actual)

PRIMARY OUTCOMES:
Causes of development of neonatal hyperbilirubinemia | 1 year
  Establish the causes contributing to the development of neonatal hyperbilirubinemia in this population, including a detailed description of the clinical course of neonates with neonatal hyperbilirubinemia.

SECONDARY OUTCOMES:
Incidence of neonatal hyperbilirubinemia | 1 year

OTHER OUTCOMES:
Clinical and biochemical risk factors for the development of neonatal hyperbilirubinemia | 1 year
Incidence of prolonged jaundice | 1 year
Neurodevelopmental outcome | 6 month
Body composition at birth, 1, 2 and 3 months of age | 3 month
Incidence of anaemia and illness episodes | 1 year
Incidence of helminthic infection | 1 year
Knowledge level and misbeliefs on neonatal hyperbilirubinemia | approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: François Nosten, Prof., Principal Investigator — Shoklo Malaria Research Unit
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Volunteers' data and results of blood sample analysis stored in our database may be shared with other researchers to use in the future. However, the other researchers will not be given any information that could identify the subject.
Supporting Information: CSR

REFERENCES:
- [Derived] Thielemans L, Trip-Hoving M, Bancone G, Turner C, Simpson JA, Hanboonkunupakarn B, van Hensbroek MB, van Rheenen P, Paw MK, Nosten F, McGready R, Carrara VI. Neonatal Hyperbilirubinemia in a Marginalized Population on the Thai-Myanmar Border: a study protocol. BMC Pediatr. 2017 Jan 21;17(1):32. doi: 10.1186/s12887-017-0798-8. PMID 28109243